CLINICAL TRIAL: NCT02004769
Title: Phase II Study of Trastuzumab in Combination With Chemotherapy (Docetaxel Plus Capecitabine) For First Line Treatment of Her2-Positive Advanced Gastric or Gastro-Esophageal Junction Cancer
Brief Title: Trastuzumab Plus Docetaxel and Capecitabine For First Line Treatment of Her2-Positive Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fudan University (Other); 307 Hospital of PLA (Other); Shandong Tumor Hospital (Other); Tongji Hospital (Other); West China Hospital (Other); Shandong Provincial Hospital (Other Government); Second Affiliated Hospital of Suzhou University (Other); Tianjin Medical University General Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Vice-president and Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28670
Record Dates: First submitted 2013-09-03; First posted 2013-12-09 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Stomach Neoplasms; Neoplasms Metastasis; ERBB2 Gene Amplification
Keywords: Metastatic gastric or gastro-esophageal junction cancer; Trastuzumab; HER2-positive; Capecitabine; Docetaxel; First-line therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab, Capecitabine, Docetaxel (Experimental): Trastuzumab(8 mg/kg loading dose followed by 6 mg/kg every 3 weeks) Capecitabine(2000mg/m2d, d1-14,every 3 weeks) Docetaxel (60mg/m2 every 3 weeks for 6 cycles).All patients will continue to receive trastuzumab and Capecitabine until either disease progression, occurrence of unacceptable toxicity or withdrawal from the study for another reason.
  Interventions: Drug: Trastuzumab; Drug: Docetaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab (Herceptin) will be administered at a loading dose of 8 mg/kg (on day 1) followed by 6mg/kg i.v. infusion every 3 weeks (q3w), until disease progress or intolerable toxicity.
  Other Names: Herceptin
Drug: Docetaxel — Docetaxel 60mg/m2 (on day 1) every 3 weeks for 6 cycles.
  Other Names: Taxotere
Drug: Capecitabine — Capecitabine (Xeloda) 2000mg/m2d, d1-14, every 3 weeks until disease progress or intolerable toxicity.
  Other Names: Xeloda

SUMMARY:
Patients with inoperable, locally advanced or recurrent and/or HER2-positive metastatic gastric or gastro-esophageal junction cancer, with no prior treatment for metastatic disease are to be recruited in the study. In the current study, the efficacy and safety of Trastuzumab in combination with Capecitabine/Docetaxel will be evaluated in Chinese patients with HER2 positive advanced or recurrent gastric cancer.60 patients could provide adequate precision rather than controlling type I&II error. Assuming the target PFS is 6.7m, 60 patients will give 90% CI of (5.5, 8.4). Considering the 5% drop out rate, 65 patients will be enrolled.

DETAILED DESCRIPTION:
This is a phase II, multi-center, open label, single arm, interventional study. Patients with HER2-positive metastatic gastric or gastro-esophageal junction adenocarcinoma who have not received prior treatment for metastatic disease will be treated with trastuzumab(8 mg/kg loading dose followed by 6 mg/kg every 3 weeks ),Capecitabine(2000mg/m2d, d1-14,every 3 weeks) and Docetaxel (60mg/m2 every 3 weeks for 6 cycles).All patients will continue to receive trastuzumab and Capecitabine until either disease progression, occurrence of unacceptable toxicity or withdrawal from the study for another reason.Primary endpoints is PFS and secondary endpoints are ORR, OS and Safety.Recruitment period:24 months;PFS follow-up period: 80% PFS events;OS follow-up period: 18 months or 80% OS events, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female. Age: 18-75 years.
2. Histologically confirmed adenocarcinoma of the stomach or gastro-esophageal junction with inoperable locally advanced or recurrent and/or metastatic disease, not amenable to curative therapy.
3. Measurable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, assessed using imaging techniques (CT or MRI).
4. HER2 positive tumor (primary tumor or metastasis, HER2 positive as defined by IHC2+ and a confirmatory FISH+ result (HER2:CEP17 ratio ≥2), or by an IHC 3+ result) as assessed by the central laboratory. Accurate and validated assay methods will be used.
5. ECOG Performance status 0-1.
6. Life expectancy of at least 3 months.
7. Signed informed consent.
8. Previous chemotherapy for advanced/metastatic disease (prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrollment into the study; adjuvant/neoadjuvant therapy with docetaxel is not allowed).

9 .Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome (e.g. patients with partial or total gastrectomy can enter the study, but not those with a jejunostomy probe).

10. Patients with active (significant or uncontrolled) gastrointestinal bleeding.

11. Residual relevant toxicity resulting from previous therapy (with the exception of alopecia), e.g. neurologic toxicity ≥ grade 2 NCI-CTCAE version 4.0.

12. Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.

13. Hematologic, Biochemical and Organ Function 14. Neutrophil count < 1.5 × 109/L, or platelet count < 100 × 109/L. 15. Serum bilirubin > 1.5 × upper limit of normal (ULN); or, AST or ALT > 2.5 × ULN (or > 5 × ULN in patients with liver metastases); or, alkaline phosphatase > 2.5 × ULN (or > 5 × ULN in patients with liver metastases, or > 10 × ULN in patients with bone but no liver metastases); or albumin < 25 g/L.

16. Creatinine clearance < 60 mL/min.

Exclusion Criteria:

1. History of documented congestive heart failure; angina pectoris requiring medication; evidence of transmural myocardial infarction on ECG; poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg); clinically significant valvular heart disease; or high risk uncontrollable arrhythmias.
2. Baseline LVEF < 50% (measured by echocardiography or MUGA).
3. Patients with dyspnea at rest due to complications of advanced malignancy or other disease, or who require supportive oxygen therapy.
4. Patients receiving chronic or high dose corticosteroid therapy. (Inhaled steroids and short courses of oral steroids for anti-emesis or as an appetite stimulant are allowed).
5. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
6. History or clinical evidence of brain metastases.
7. Serious uncontrolled systemic intercurrent illness, e.g. infections or poorly controlled diabetes.
8. Positive serum pregnancy test in women of childbearing potential.
9. Subjects with reproductive potential not willing to use an effective method of contraception.
10. Received any investigational drug treatment within 4 weeks of start of study treatment.
11. Radiotherapy within 4 weeks of start of study treatment (2 week interval allowed if palliative radiotherapy given to bone metastatic site peripherally and patient recovered from any acute toxicity).
12. Major surgery within 4 weeks of start of study treatment, without complete recovery.
13. Patients with known active infection with HIV, HBV, or HCV.
14. Known hypersensitivity to any of the study drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
PFS(Progression-free survival ) | up to 4 years
  The PFS was calculated from the initiation of chemotherapy to the date of disease progression or death,

SECONDARY OUTCOMES:
ORR (Overall tumor response) | up to 4 years
  Overall tumor response: This is defined as the occurrence of either a confirmed complete (CR) or a partial (PR) best overall response as determined by the RECIST criteria from confirmed radiographic evaluations of target and non-target lesions.
OS (Overall survival ) | up to 4 years
  Overall survival was measured from the initiation of chemotherapy to the date of the last follow-up or death.
Safety | up to 4 years
  Adverse events and laboratory tests graded according to the NCI-CTC AE Version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, M.D,Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sawada N, Ishikawa T, Fukase Y, Nishida M, Yoshikubo T, Ishitsuka H. Induction of thymidine phosphorylase activity and enhancement of capecitabine efficacy by taxol/taxotere in human cancer xenografts. Clin Cancer Res. 1998 Apr;4(4):1013-9. PMID 9563897
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Background] Roth AD, Fazio N, Stupp R, Falk S, Bernhard J, Saletti P, Koberle D, Borner MM, Rufibach K, Maibach R, Wernli M, Leslie M, Glynne-Jones R, Widmer L, Seymour M, de Braud F; Swiss Group for Clinical Cancer Research. Docetaxel, cisplatin, and fluorouracil; docetaxel and cisplatin; and epirubicin, cisplatin, and fluorouracil as systemic treatment for advanced gastric carcinoma: a randomized phase II trial of the Swiss Group for Clinical Cancer Research. J Clin Oncol. 2007 Aug 1;25(22):3217-23. doi: 10.1200/JCO.2006.08.0135. PMID 17664469
- [Background] Thuss-Patience PC, Kretzschmar A, Repp M, Kingreen D, Hennesser D, Micheel S, Pink D, Scholz C, Dorken B, Reichardt P. Docetaxel and continuous-infusion fluorouracil versus epirubicin, cisplatin, and fluorouracil for advanced gastric adenocarcinoma: a randomized phase II study. J Clin Oncol. 2005 Jan 20;23(3):494-501. doi: 10.1200/JCO.2005.02.163. PMID 15659494